CLINICAL TRIAL: NCT00919581
Title: Pilot Study: The Role of Macrophage Migration Inhibitory Factor (MIF) in Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Ona Bloom, Associate Professor, Northwell Health
Other Study IDs: 0268
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy controls
- Subjects with spinal cord injury

SUMMARY:
The purpose of the study is to investigate inflammatory and other substances that may be elevated in the blood and blood cells following spinal cord injury (SCI). These substances will be evaluated in samples from people who have had a spinal cord injury due to trauma (e.g. car accident or a fall) within the first week (acute) or at least one year ago (chronic). Specifically, the study will evaluate the presence and levels of a protein, macrophage migration inhibitory factor (MIF). MIF is released by cells and has a specific effect on the way cells behave, communicate and work together. In several other medical conditions, MIF is known to increase inflammation in the body. By comparing blood samples from individuals with spinal cord injury and uninjured (no spinal cord injury) individuals, the investigators will try to find out if MIF levels are increased in people with SCI. Investigators will also use these samples to measure other proteins that increase inflammation in the body and to see if the biological activities of MIF can be reduced in a test tube by adding other substances to the blood samples. It is hoped that this study of MIF and other proteins related to inflammation will help improve the treatment of SCI in the future.

We hope to enroll a total of 312 subjects in this study (50 with acute spinal cord injury, 125 with chronic spinal cord injury, and 137 uninjured individuals).

DETAILED DESCRIPTION:
During the study visit the investigator will collect basic biographical information and health information, including some questionnaires, from the subjects and their medical record.

Acute SCI subjects will also have blood drawn once daily (First blood draw will approximately be 2 tablespoons and subsequent blood draws will approximately be 1 tablespoon) .

Chronic SCI subjects will have blood drawn per study visit (approximately 2 tablespoons) and will be asked to participate in two study visits, to take place 6 months apart.

ELIGIBILITY:
Inclusion Criteria:

SCI Subject Inclusion Criteria: To be eligible for prospective enrollment, subjects are required to meet the following inclusion criteria:

* ≥18 years of age
* History SCI (acute or chronic): All American Spinal Injury Association (ASIA) classifications A-D and all levels.

Healthy Control Subject Inclusion Criteria: To be eligible for prospective enrollment, healthy control subjects are required to meet the following inclusion criteria:

* ≥18 years of age
* The absence of any current or previous medical conditions

To be eligible for prospective enrollment, SCI subjects are required to not meet the following exclusion criteria:

* < 18 years of age
* No known SCI
* Concurrent infection such as UTI
* Deep pressure sores
* cancer, chemotherapy or neutropenia
* autoimmune disease

Healthy Control Subject Exclusion Criteria: To be eligible for prospective enrollment, healthy control subjects are required to not meet the following exclusion criteria:

* < 18 years of age
* Current or previous medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with spinal cord injury, uninjured controls
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2009-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
MIF | 2
  macrophage migration inhibitory factor (MIF), a pro-inflammatory cytokine

SECONDARY OUTCOMES:
inflammatory mediators | 2
  circulating inflammatory mediators

CONTACTS AND LOCATIONS:
Overall Officials: Ona Bloom, PhD, Principal Investigator — Northwell Health
Locations (1):
- Feinstein Institute for Medical Research, Northwell Health, Manhasset, New York, United States

REFERENCES:
- [Background] Bank M, Stein A, Sison C, Glazer A, Jassal N, McCarthy D, Shatzer M, Hahn B, Chugh R, Davies P, Bloom O. Elevated circulating levels of the pro-inflammatory cytokine macrophage migration inhibitory factor in individuals with acute spinal cord injury. Arch Phys Med Rehabil. 2015 Apr;96(4):633-44. doi: 10.1016/j.apmr.2014.10.021. Epub 2014 Nov 15. PMID 25461821
- [Result] Stein A, Panjwani A, Sison C, Rosen L, Chugh R, Metz C, Bank M, Bloom O. Pilot study: elevated circulating levels of the proinflammatory cytokine macrophage migration inhibitory factor in patients with chronic spinal cord injury. Arch Phys Med Rehabil. 2013 Aug;94(8):1498-507. doi: 10.1016/j.apmr.2013.04.004. Epub 2013 Apr 22. PMID 23618747